CLINICAL TRIAL: NCT04679571
Title: Efficacy of Targeted And Response-Guided Albumin Therapy Versus Standard Medical Treatment In Outcomes Of Recurrent Ascites In Patients With Decompensated Cirrhosis- A Randomized Controlled Trial".
Brief Title: Efficacy of Targeted And Response-Guided Albumin Therapy Versus Standard Medical Treatment In Outcomes Of Recurrent Ascites In Patients With Decompensated Cirrhosis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-38
Record Dates: First submitted 2020-10-27; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-08

CONDITIONS: Decompensated Cirrhosis
MeSH Terms: interventions — Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted Albumin with Standard Medical Treatment (Experimental): Patients with serum albumin <3 g/L with recurrent ascites - Will receive 20 % albumin at 60 grams/week until target serum albumin of 3.0 g/L is achieved following this patients would get 40 grams of albumin every week until ascites resolution or serum albumin >3.5 g/L. Patients who achieve this target will continue with 20 gm/week until patient has complete resolution of ascites and serum albumin >3.5 gm/L this patients would receive albumin 20 gms once every 2 weeks
  Interventions: Biological: Albumin; Drug: Standard Medical Treatment
- Standard Medical Treatment (Active Comparator): Standard Medical Treatment- Salt-restriction, diuretics with large volume paracentesis These patients will be put on low sodium diet (2 g/day) and will be given a combination of loop diuretic (furosemide 40-160 mg/day) and a distal acting diuretic (spironolactone 100-400 mg/day) with dose escalation by one step at a time with monitoring for side-effects. Large volume paracentesis (LVP) will be performed along with intravenous albumin (8 g/L ascites removed) as required with record of the frequency of taps.
  Follow up: 2 week, 4 weeks then every 3 months for 1 year
  Interventions: Drug: Standard Medical Treatment

INTERVENTIONS:
Biological: Albumin — Patients with serum albumin <3 g/L with recurrent ascites - Will receive 20 % albumin at 60 grams/week until target serum albumin of 3.0 g/L is achieved following this patients would get 40 grams of albumin every week until ascites resolution or serum albumin >3.5 g/L. Patients who achieve this target will continue with 20 gm/week until patient has complete resolution of ascites and serum albumin >3.5 gm/L this patients would receive albumin 20 gms once every 2 weeks.
  Arms: Targeted Albumin with Standard Medical Treatment
Drug: Standard Medical Treatment — Standard Medical Treatment- Salt-restriction, diuretics with large volume paracentesis These patients will be put on low sodium diet (2 g/day) and will be given a combination of loop diuretic (furosemide 40-160 mg/day) and a distal acting diuretic (spironolactone 100-400 mg/day) with dose escalation by one step at a time with monitoring for side-effects. Large volume paracentesis (LVP) will be performed along with intravenous albumin (8 g/L ascites removed) as required with record of the frequency of taps.
  Follow up: 2 week, 4 weeks then every 3 months for 1 year.

SUMMARY:
The current prospective randomized controlled trial would aim to study the efficacy of targeted albumin therapy versus standard medical treatment in reduction in 6-month mortality in recurrent ascites in patients with decompensated cirrhosis. Additionally, we aim to evaluate the efficacy of albumin in decreasing the incidence of complications: paracentesis induced circulatory dysfunction (PICD), AKI, hyponatremia, bacterial infections, hepatic encephalopathy and variceal bleed, impact on systemic hemodynamics and portal pressures, renal reserve as assessed by biomarkers and on immunomodulation. In this open labeled randomized study, consecutive cirrhotic patients, fulfilling the inclusion criteria and exclusion criteria will be enrolled in the study.

The patients will be randomized to 2 groups by the clinical trial coordinator (CTC). The CTC will be blind to the patient and treatment received, and the allocation concealment by the sequentially numbered opaque sealed envelopes (SNOSE) technique would be done. Patients would be assessed every 2 weeks for first 8 weeks with serum albumin levels, ascites grade and use of diuretics and then every 3 months. The treatment would receive targeted albumin therapy as detailed in methods while patients in the other group would receive standard medical treatment. The primary outcome of the study would be evaluation of 6-month mortality while secondary outcome measures would be the incidence of liver-related complications at 3, 6 and 12 months, survival free of liver transplant and TIPS in both groups at 6 months and 1 year, improvement in quality of Life as assessed by short form survey-36 version (SF-36) at 6 and 12 months, improvement in renal reserve (as assessed by renal biomarkers) at 3, 6 and 12 months, reduction in the frequency of large volume paracentesis at 3, 6 and 12 months and change in immune parameters at 3 and 6 months.

DETAILED DESCRIPTION:
Study Design Aim & Objectives Primary

• To study the efficacy of targeted albumin therapy versus standard medical treatment in reduction in 6-month mortality in recurrent ascites in patients with decompensated cirrhosis

Secondary Objectives

* To study the frequency of therapeutic paracentesis in both groups
* Incidence of complications: paracentesis induced circulatory dysfunction (PICD), AKI, hyponatremia, bacterial infections, hepatic encephalopathy and variceal bleed
* Impact on systemic hemodynamics and portal pressures
* Impact on fraility and sarcopenia
* Time to resolution of ascites in both groups
* Changes in renal reserve as assessed by sequential Cystatin C based equations for eGFR and other biomarkers (urine-NGAL, Kidney Injury molecule-1, Liver-Fatty Acid Binding Protein (L-FABP) every 3 months)
* Adverse effects and discontinuation rates of beta-blockers in both groups
* Survival free of liver transplant and TIPS in both groups at 6 months and 1 year
* Quality of Life as assessed by short form survey-36 version (SF-36)
* Effect of albumin therapy on immunomodulation
* Effect of albumin on 12-month mortality

Methodology DOSING REGIMEN (Describe the subject or animal dosing) In this open labeled randomized study, consecutive cirrhotic patients, fulfilling the inclusion criteria and exclusion criteria will be enrolled in the study. Details of sample size calculation are given under section of statistical methods. Severity of liver disease will be assessed according to severity scores- CTP and MELD score.

The patients will be randomized to 2 groups by the clinical trial coordinator (CTC). The CTC will be blind to the patient and treatment received, and the allocation concealment by the sequentially numbered opaque sealed envelopes (SNOSE) technique would be done. Patients would be assessed at 2 weeks, 4 weeks with serum albumin levels, ascites grade and use of diuretics and then every 3 months

Group A- Would receive standard medical treatment (details as in patients for Group B) plus Targeted albumin therapy would be given as under:

Patients with serum albumin <3 g/L with recurrent ascites - Will receive 20 % albumin at 60 grams/week until target serum albumin of 3.0 g/L is achieved following this patients would get 40 grams of albumin every week until ascites resolution or serum albumin >3.5 g/L. Patients who achieve this target will continue with 20 gm/week until patient has complete resolution of ascites and serum albumin >3.5 gm/L or a maximum of 6 months following this patients would receive albumin 20 gms once every 2 weeks Group B: Standard Medical Treatment- Salt-restriction, diuretics with large volume paracentesis These patients will be put on low sodium diet (2 g/day) and will be given a combination of loop diuretic (furosemide 40-160 mg/day) and a distal acting diuretic (spironolactone 100-400 mg/day) with dose escalation by one step at a time with monitoring for side-effects. Large volume paracentesis (LVP) will be performed along with intravenous albumin (8 g/L ascites removed) as required with record of the frequency of taps.

Follow up: 2 week, 4 weeks then every 3 months for 1 year

Important definitions:

Recurrent ascites will be defined as ascites that recurs on at least three occasions within a 12-month period despite dietary sodium restriction and adequate diuretic doses.

Ascites resolution would be defined as absence of clinical ascites (ascites grade 0 or 1) which can either be partial- Would be defined as resolution of ascites on diuretics and complete would be defined as resolution of ascites without the need of diuretics.

Investigations: Baseline HVPG with assessment of portal (systemic and pulmonary hemodynamics) and cardiac hemodynamics, cystatin C, plain CT scan for assessment of sarcopenia. Body weight, blood pressure and echocardiogram would be done for all patients. Glomerular filtration rate (GFR) will be estimated by using eGFR equations -modification of diet in renal disease (MDRD6) and Cystatin C based (Chronic kidney disease Epidemiology Collaboration). Along with this, arterial blood sample will be collected after overnight fast and bed rest at least for 8 h in supine position for plasma renin activity, plasma aldosterone and plasma norepinephrine concentration. A baseline urinalysis with assessment of urinary sodium would also be done for all enrolled patients. Patients would subsequently undergo HVPG after 3-6 months and cystatin C every 3 months. Apart from this, urine neutrophil-gelatinase associated lipocalin (NGAL), plasma renin activity and serum aldosterone levels would be performed at baseline, 3 and 6 months. A repeat plain CT scan to assess sarcopenia would be done at 3 months and at 6 months. The follow up would be 1 year or until TIPS or liver transplant.

Albumin related immunological assessment:

Considering immunomodulation as an important mechanism of action of albumin. Additional experiments would be done at baseline, 3 and 6 months to assess the albumin isoforms (HMA, HNA1, HNA2, IMA) , levels of pro-inflammatory and anti-inflammatory cytokines (multiplex luminex based cytokine array) , inflammatory mediators (C-Reactive Protein, endotoxin assay, compliment proteins; DAMPS ); Frequency and functional profile of innate immune cells (monocytes, neutrophills)

Albumin isoforms analysis:

Chemicals Change in albumin isoform will be done by quantification of different albumin modification(HMA, HNA1, HNA2, IMA) on an electron spray ionization orbitrap HRMS system "(Q Exative plus) mass spectrometer coupled to UHPLC from Thermoscientific USA.Briefly the isolated plasma of patients blood at given time point (day 0 and three month) will be diluted with distilled water at a 1:4,000 ratio, and then 8 uL of this diluted plasma will be injected into the high performance liquid chromatography-electron spray ionization MS system. High-performance liquid chromatography separation will be performed on a reverse-phase C8 column (Agilent ZORBAX RRHD 300SB-C8, 2.1 mm id 3 50 mm, 1.8 lm threaded column with a pore size of 300 Å) at a flow rate of 0.2 mL/minute using an H2O-acetonitrile (with 0.1% formic acid) solvent system under a gradient of 90% H2O to 90% acetonitrile over a period of 25 minutes with acquisition starting at 3 minutes. Under auto-MS conditions, mass spectral analysis will be performed. A similar analysis will also be performed with exogenous albumin solution. The obtained compound electron spray ionization MS spectra will be analyzed using the software Protein Deconvolution soft warre (thermoscientific germany). Here, after minimizing the base peak chromatogram from the total ion chromatogram, albumin mass chromatograms will be obtained and analyzed. The obtained albumin spectra will then be deconvoluted within mass range from 66,000-67,000 Da (as the molecular weight [MW] of various albumin isoforms fall within this range. Finally, from the intensity of the peaks, the abundance of albumin isoforms will be measured and the relative abundance of the various HSA isoforms will be reported as described in Das et.al 2017. This will be performed at baseline and 3 months. ( Mass spectrometry (MS)-grade water, acetonitrile, and formic acid will be purchased from Sigma-Aldrich (St. Louis, MO). Purified HSA was purchased from Baxter (Gurgaon, India). All reagents will be of analytical grade.

Cytokine array A panel of 45 cytokines, chemokines, and growth factors will be analyzed in blood plasma of patients group at baseline and 3 months using a Bio-Plex multiplex cytokine bead assay system (Bio-Rad, CA) as per the manufacturer's protocol. The intra-assay and inter assay coefficient of variation considered for multiplex assays will be < 5%

Innate Immune cells profiling:

Total whole blood will be collected from patients pre and post therapy and evaluated for % frequency of monocytes by staining with fluorochrome labeled anti-CD14 anti CD16 and for neutrophils anti-CD11b anti CD16 anti-CD15, anti-CD66b and will acquired and anlaysed using flow cytometry FACS verse (BD biosciences). For the functional profiling of innate immune cells, the blood will be divided into two parts. The PBMCs will be isolated using ficoll-hypaque (Himedia) and monocytes will be isolated using CD14 isolation kit from miltenyi biotech as per the manufacture protocol. Whereas, other part of the blood will be used to isolate the neutrophils using gran-hypaque (Himedia). The intracellular cytokines such as IFN-y, TNF-a, IL-1b will be analysed after low dose of LPS stimulation. Also, phagocytic burst or ROS generation will be done using manufacturer's described protocol. Again the data will be acquired and anlysed using FACS verse (BD biosciences).

Seahorse metabolic analysis methodology:

Effect on energy metabolism of monocytes (that guide the functional property of immune cells) we be analyzed by measuring the extracellular acidification rate (ECAR) and oxygen consumption rate (OCR) through Seahorse XF24 Extracellular Flux Analyzer instrument in peripheral blood monocytes of patients at baseline and 3 months as a measure of lactate production (a surrogate for the glycolytic rate) and OXPHOS respectively. In brief, monocytes will be isolated from freshly collected blood using CD14 isolation kit from miltenyi biotech as per the manufacture protocol. Isolated monocytes will be seeded in triplicate at a density of 1X105 cells per well. Prior to starting the assay, cells will be incubated in Seahorse Assay Medium supplemented with 10 mM glucose and 1 mM sodium pyruvate and glutamine in 37°C incubator without CO2 for 45 min. Further change in parameters of oxidative phosphorylation will be calculated by a real-time change in OCR in response to treatment with Oligomycin (ATPase inhibitor, 1 μM), FCCP (0.2 μM) and rotenone (0.5 μM).

Study Population:

SUBJECT POPULATION/PRE-CLINICAL MODEL (Describe the subject population including inclusion/exclusion criteria or animal model)

Study Design:

* A randomized controlled study.
* The study will be conducted on patients admitted to Department of Hepatology from August 2020 to August 2022 at ILBS, New Delhi
* Study group will comprise of patients of decompensated cirrhosis with recurrent ascites

Sample Size calculation: In the randomized controlled trial by Singh et al (Journal of Hepatology 2012) the 90-day mortality in patients of recurrent ascites on midodrine was 15/20 (75%) vs. 8/20(40% ) in the standard medical treatment group (large volume paracentesis and albumin infusions). Assuming that the survival for albumin is 75% and with SMT is 40%, then with alpha of 5% and power 90% we need to enroll 90 cases i.e 45 cases in each group. Further assuming 10% drop out rate we need to enroll 100 cases 50 each group and randomly allocated with block randomisation method with block size taken as 10.

Proportion of survival in the treatment group at a given time point = 0.75 Proportion of survival in the control group at a given time point = 0.40 Hazard ratio = 3.19 Power (%) = 90 Alpha Error (%) = 5 Sided = 2 Required sample size for treatment group = 45 Required sample size for control group = 45 Alpha Error (%) Power (%) First Group Second Group 5 70 27 27 80 34 34 90 45 45

Intervention: Targeted albumin therapy Monitoring and Assessment: Follow up: 2 weeks, 4 weeks, 3 months, then every 3 months for 1 year

Statistical analysis

* All variables shall be expressed in mean (sd) or median (range)
* Variables will be compared by Mann- Whitney U test
* For Categorical variables we will use Chi-Square or Fisher's test
* Survival analysis will be done using Cox-proportional regression analysis
* Actuarial probability of survival shall be calculated by Kaplan- Meier graph and compared by log- rank test.
* Competing risk survival analysis with competing events as TIPS and liver transplant would be performed Adverse Effects: Allergic reactions to albumin, worsening of dyspnea, volume overload Stopping rule: Reaction to albumin infusion

Ethical issues in the study and plans to address these issues:

There are no ethical issues with respect to the trial protocol. Albumin is routinely recommended for the management of patients with cirrhosis with ascites. In a large multicentric trial it was shown that high dose of albumin of 40 grams/week improved outcomes in cirrhotics with uncomplicated ascites. This however lacks clinical application based on feasibility to provide high doses in a resource constraint country like India. Our data would therefore provide a targeted approach (escalation/de-escalation) based on response individualised for each patient and its effect on imrpving overall outcomes. The study drug would be provided free of cost and the cost of special investigations which are not part of the standard of care would not be borne by the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cirrhosis of liver with recurrent ascites.
2. Patients with age from 18-70 years

Exclusion Criteria:

1. Renal failure (Creatinine >1.5mg/dl)
2. Recent Gastrointestinal bleeding within 7 days
3. Spontaneous bacterial Peritonitis
4. Patients with organic nephropathy ( as defined by IAC)
5. Patients with Cardiovascular disease or chronic obstructive pulmonary disease
6. Systemic arterial hypertension (>160/90mmhg)
7. Presence of hepatocellular carcinoma (outside Milan criteria)( or portal vein thrombosis
8. Budd-Chiari Syndrome
9. Patients with active sepsis
10. Pregnancy
11. Patients with hepatic encephalopathy
12. No use of drugs affecting systemic hemodynamics 7 days prior to enrolment (except beta-blockers)
13. Patients with serum albumin >3 gm
14. Refusal to participate
15. Known or suspected hypersensitivity to albumin
16. Prior TIPS
17. Post liver or kidney transplantation
18. Patients enrolled in other clinical trials
19. Extrahepatic malignancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-30 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Mortality in both groups | 6 months

SECONDARY OUTCOMES:
Incidence of liver-related complications in both groups | 3 months
Incidence of liver-related complications in both groups | 6 months
Incidence of liver-related complications in both groups | 12 months
Survival free of liver transplant in both groups | 6 months
Survival free of liver transplant in both groups | 12 months
Number of patients underwent TIPS (Transjugular Intrahepatic Portosystemic Shunt) in both groups | 6 months
Number of patients underwent TIPS (Transjugular Intrahepatic Portosystemic Shunt) in both groups | 12 months
Change in quality of Life as assessed by short form survey-36 version (SF-36) in both groups | 6 months
Change in quality of Life as assessed by short form survey-36 version (SF-36) in both groups | 12 months
Change in renal reserve (as assessed by renal biomarkers) in both groups | 3 months
  urine NGAL, CYSTATIN C AND KIM1 will be done
Change in renal reserve (as assessed by renal biomarkers) in both groups | 6 months
  urine NGAL, CYSTATIN C AND KIM1 will be done
Change in renal reserve (as assessed by renal biomarkers) in both groups | 12 months
  urine NGAL, CYSTATIN C AND KIM1 will be done
Change in the frequency of large volume paracentesis in both groups | 3 months
Change in the frequency of large volume paracentesis in both groups | 6 months
Change in the frequency of large volume paracentesis in both groups | 12 months
Improvement in pro inflammatory cytokines | 3 months
  TNF ALPHA, IL6, CRP AND IL1BETA will be done
Improvement in pro inflammatory cytokines | 6 months
  TNF ALPHA, IL6, CRP AND IL1BETA will be done
Mortality in both groups | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India